CLINICAL TRIAL: NCT06926439
Title: Prediction of Detoxification Effect of Fat Emulsion Based on Drug Diffusion Law: Clinical Observational Study
Brief Title: Prediction of Detoxification Effect of Fat Emulsion Based on Drug Diffusion Law
Status: Active, not recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, MD, PhD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2024-LCYJ-MS-06; 2024-LCYJ-MS-06 (Other Grant/Funding Number: Nanjing Drum Tower Hospital)
Record Dates: First submitted 2025-01-23; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Poisoning; Toxicokinetics; Lipid Emulsion
MeSH Terms: conditions — Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — plasma

INTERVENTIONS:
Drug: Long chain lipid emulsion — For patients presenting with fat soluble drug overdose, administer a weight-based infusion of long-chain lipid emulsion at 0.05 ml/kg/min for 1 hour, not to exceed a total of 250 mL.

SUMMARY:
The goal of this observational study is to establish a predictive model for the clinical use value of fat emulsion as an antidote based on the physical information of fat emulsion on drug diffusion process.

The main question it aims to answer is:

Observing the effect of fat emulsion on the pharmacokinetic changes of overdose drugs; Observe and evaluate the therapeutic effect of long-chain fat emulsion as an antidote; Participants will have their whole blood samples collected for toxicology testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clear history of acute drug exposure;
* The exposed drug is a lipid soluble drug (with a lipid water distribution coefficient logP>0);
* Age: 18-85 years old;
* The patient or guardian agrees to participate in this project and signs an informed consent form;

Exclusion Criteria:

* Patients with shock and severe lipid metabolism disorders (such as hyperlipidemia);
* Patients with unclear exposure history;
* Drug exposure time > 24 hours;
* Exposure to two or more drugs;
* Select patients with specific detoxifying agents;
* Merge patients with severe cardiovascular and cerebrovascular diseases;
* Patients with negative blood toxicity test results or overdose of non-fat-soluble drugs;
* Those who fail to provide complete general information and clinical data;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department of Nanjing Drum Tower Hospital admits patients
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of the Overdosed Drug | From baseline (pre-emulsion infusion) up to 24 hours post-infusion
  The highest observed plasma concentration of the overdosed drug following administration of long-chain lipid emulsion. Blood samples will be collected at predefined intervals to quantify drug concentration and assess the impact of fat emulsion on peak levels.
Time to Maximum Plasma Concentration (Tmax) of the Overdosed Drug | From baseline (pre-emulsion infusion) up to 24 hours post-infusion
  The time point at which the plasma concentration of the overdosed drug reaches its maximum level. This will help determine whether long-chain lipid emulsion alters the rate of drug absorption or distribution.
Area Under the Plasma Concentration-Time Curve From 0 to Last Measurable Concentration (AUC0-last) | From baseline (pre-emulsion infusion) up to 24 hours post-infusion
  The area under the plasma concentration-time curve from time 0 to the last measurable concentration. This is used to evaluate the overall drug exposure and how it may be modified by the fat emulsion.
Terminal Elimination Half-Life (t½) of the Overdosed Drug | From baseline (pre-emulsion infusion) up to 24 hours post-infusion
  The time required for the plasma concentration of the overdosed drug to decrease by half. This measure will be used to assess whether long-chain lipid emulsion accelerates drug clearance.
Plasma Clearance (CL) of the Overdosed Drug | From baseline (pre-emulsion infusion) up to 24 hours post-infusion
  The volume of plasma completely cleared of the overdosed drug per unit time, assessing how fat emulsion influences the drug's elimination.
Elimination Rate Constant (Ke) of the Overdosed Drug | From baseline (pre-emulsion infusion) up to 24 hours post-infusion
  The first-order elimination rate constant indicating the speed at which the drug is removed from the body, measured using plasma concentration data over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China